CLINICAL TRIAL: NCT01402843
Title: A Randomized, Double Blind, Double Dummy, Placebo Controlled Phase III Trial to Evaluate the Efficacy, Safety of Coadministered Pitavastatin and Valsartan in Patients With Hypertension and Dyslipidemia(COCTAIL Study)
Brief Title: Efficacy, Safety of Coadministered Pitavastatin and Valsartan in Patients With Hypertension and Dyslipidemia
Acronym: COCTAIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Gyu Rok Han / MD, Hallym University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CWP-PTV-301
Record Dates: First submitted 2011-07-14; First posted 2011-07-26 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension; Dyslipidemia
Keywords: phase III combination study
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — pitavastatin; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- pitavastatin + valsartan (Experimental)
  Interventions: Drug: pitavastatin, valsartan, placebo
- pitavastatin + placebo (Placebo Comparator)
  Interventions: Drug: pitavastatin, valsartan, placebo
- valsartan + placebo (Placebo Comparator)
  Interventions: Drug: pitavastatin, valsartan, placebo
- placebo (Placebo Comparator)
  Interventions: Drug: pitavastatin, valsartan, placebo

INTERVENTIONS:
Drug: pitavastatin, valsartan, placebo — pitavastatin 4mg/day 8 week valsartan 320mg/day 8 week
  Other Names: Livalo, Diovan

SUMMARY:
Pitavastatin, a representative statin-series anti-dyslipidemic drug, and Valsartan, a representative ARB-series anti-hypertensive drug, have been authorized for use also in South Korea. They have been tested in many countries and proved to be effective and safe. The concurrence of dyslipidemia and hypertension has a higher rate, hence statin-series drugs and antihypertensive drugs are simultaneously administered to such patients. The combined administration of statin-series drugs and CCB-series drugs have.

DETAILED DESCRIPTION:
This clinical trial was conducted to evaluate the safety and effectiveness of the combined administration of Pitavastatin and Valsartan to ethnic Koreans with dyslipidemia concurrent with hypertension, as well as to research the influence on the pharmacodynamic interaction between the two drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 and older
2. Patients with Dyslipidemia
3. Patients with hypertension
4. Patients who voluntarily signed the consent form.

Exclusion Criteria:

1. Blood Pressure

   * In case there is a sitting systolic blood pressure difference of 20mmHg and over or sitting diastolic blood pressure is 10mmHg and over in selected arm.
   * Patients with symptomatic orthostatic hypotension.
   * Patients having the history of Secondary hypertension or suspected to be Secondary hypertension, e.g., aortic coarctation, hyperaldosteronism, renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic renal disease, etc.
2. Patients with severe heart diseases (NYHA class-III and IV), with ischemic heart diseases (angina pectoris and myocardial infarction) and with peripheral vascular diseases, and patients who underwent percutaneous transluminal coronary angioplasty (PTCA) or treatments for coronary artery bypass graft within 6 months.
3. Patients with clinically significant ventricular tachycardia or atrial fibrillation or atrial flutter, and patients with arrhythmia judged to be clinically significant by investigators.
4. Patients with hypertrophic obstructive cardiomyopathy, severe obstructive CAD, aortic stenosis and hemodynamically significant aortostenosis or mitral stenosis.
5. Patients with severe cerebrovascular diseases.
6. Patients with severe or malignant retinosis.
7. Patients with consumption diseases or autoimmune diseases or connective tissue diseases
8. Patients with endocrine or metabolic diseases that are known to affect serum lipid or lipoprotein.

   * Patients with uncontrollable diabetes
   * Patients with uncontrollable thyroid dysfunction
9. Patients who underwent treatments that may affect lipid before the clinical trial.
10. Patients having the history of myopathy or rhabdomyolysis.
11. Patients with severe renal disorders or hepatic disorders.
12. Patients with gastrointestinal diseases that may affect drug absorption, distribution, metabolism and excretion or who underwent such operations, or patients with present active gastritis or gastrointestinal hemorrhage or proctorrhagia or active and inflammatory bowel syndrome that has occurred within 12 months.
13. All of patients with chronic inflammatory diseases whereto anti-inflammatory treatments need to be applied.
14. Patients having the history of drug or alcohol abuse.
15. Pregnant women and/or women in the lactation period or the child-bearing period.
16. Patients who are hypersensitive to Pitavastatin and Valsartan.
17. Patients who have taken other investigational drugs within 3 months before undergoing the screening test for this clinical trial.
18. Patients judged to be unsuitable for this clinical trial by investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The experimental group should be compared with control group in the change of DBP and LDL-C on the basis of the baseline. | 8 week

SECONDARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure at 6 months. | 8 week
The changes and rate of lipid variables (TG, TC, HDL cholesterol and apolipoprotein B) | 8 week

CONTACTS AND LOCATIONS:
Overall Officials: Gyu Rok Han, MD, Principal Investigator — Dept. of Cardiology, Hallym University Medical Center
Locations (10):
- South Korea (10):
  - Chungbuk National University Hospital, Chungju
  - Konyang University Hospital, Daejeon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Ajou University Medical Center, Suwon